CLINICAL TRIAL: NCT01146184
Title: Single Incision Laparoscopic Cholecystectomy Using a Flexible Endoscope and Ethicon Manually Articulating Devices (MAD)
Acronym: IRB#08-181
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: the manufacturer never released the instruments
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 08-181
Record Dates: First submitted 2010-06-01; First posted 2010-06-17 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2015-08

CONDITIONS: Cholelithiasis; Pain
Keywords: Cholelithiasis; Single Incision; Flexible Endoscope; Ethicon Manually Articulating Device; Pain
MeSH Terms: conditions — Cholelithiasis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-Incision Cholecystectomy (Experimental): Extracting the gallbladder laparoscopically is made difficult through a single incision.
  Interventions: Device: Flexible endoscope and Ethicon Manually Articulating Device

INTERVENTIONS:
Device: Flexible endoscope and Ethicon Manually Articulating Device — Using the Flexible Endoscope and the Ethicon Manually Articulating Device, removal of the gallbladder through a single incision is improved.
  Other Names: Single Incision cholecystectomy using flexible endoscope; Ethicon instruments

SUMMARY:
The aim of this study is to improve the technique of laparoscopic cholecystectomy by using a flexible endoscope passed through a single umbilical skin incision, as previously reported, now with the use of Manually Articulating Devices (Ethicon Endo-Surgery, Inc.) through the endoscope.

DETAILED DESCRIPTION:
Single incision laparoscopic surgeries (SILS) have taken a step further the field of minimally invasive surgery with reports of a variety of laparoscopic procedures performed through a single incision.

However the technique is challenging due to the proximity of the instruments passed through the single umbilical skin incision. Several improvisions were made to accommodate this technical restriction by making flexible umbilical ports that accommodate several trocars, or usage of different length instruments to strategically place the surgeons, minimizing collision and improving ergonomics.

The flexibility of the endoscope will allow improved freedom of movement within the abdominal cavity and ease of gallbladder dissection. The investigators believe that this technique will take advantage of the flexible nature of the endoscope while avoiding the risks of transluminal surgery inherent in natural orifice surgery. Flexible endoscope offers an excellent solution to SILS, with its flexible optics and ability to pass working instruments through it.

The flexible endoscope to be used ia a 12mm dual channel Karl Storz or Olympus gastroscope.Ethicon instruments are essentially like traditional endoscopic instruments with an extra joint at the working end, mimicking a wrist joint. These instruments are FDA listed/cleared pursuant to 510(k) provisions of the Food, Drug and Cosmetic Act with general indications for use in endoscopic or laparoscopic procedures. We will be using an articulating grasper, articulating biopsy forcepts, and an articulating needle knife.

We will measure pain with pain scales.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated Biliary Colic
* ASA I or II

Exclusion Criteria:

* Pregnant Women
* Children
* Institutionalized mentally disabled
* Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Improving the technique of laparoscopic Cholecystectomy with Flexible Endoscope and Ethicon Manually Articulating Device | Intra-Operative
  Using flexible endoscopes and the Ethicon Manually Articulating Device will facilitate the procedure of removing the gallbladder by allowing more flexibility and greater movement in the abdominal cavity, better triangulation for dissection and increased quality of optics for the single-incision technique.

SECONDARY OUTCOMES:
Post-operative Pain | 1 month
  Single-Incision laparoscopic cholecystectomy to reduce pain, improve patient outcomes and minimize invasiveness.
Complications | 1 month
  Measure intra-operative and post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Julio Teixeira, MD, Principal Investigator — St Luke's Roosevelt Hospital Center- Surgery Department
Locations (1):
- St Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Background] Ng WT, Kong CK, Wong YT. One-wound laparoscopic cholecystectomy. Br J Surg. 1997 Nov;84(11):1627. No abstract available. PMID 9393287
- [Background] Teixeira J, McGill K, Koshy N, McGinty J, Todd G. Laparoscopic single-site surgery for placement of adjustable gastric band--a series of 22 cases. Surg Obes Relat Dis. 2010 Jan-Feb;6(1):41-5. doi: 10.1016/j.soard.2009.03.220. Epub 2009 Apr 16. PMID 19560980
- [Background] Petersen LR, Doll LS. Human immunodeficiency virus type 1-infected blood donors: epidemiologic, laboratory, and donation characteristics. The HIV Blood Donor Study Group. Transfusion. 1991 Oct;31(8):698-703. doi: 10.1046/j.1537-2995.1991.31892023493.x. PMID 1926312
- [Background] Slim K, Pezet D, Stencl J Jr, Lechner C, Le Roux S, Lointier P, Chipponi J. Laparoscopic cholecystectomy: an original three-trocar technique. World J Surg. 1995 May-Jun;19(3):394-7. doi: 10.1007/BF00299168. PMID 7638995